CLINICAL TRIAL: NCT03627312
Title: Omega-3 Supplements to Reduce Antisocial Behaviour in Young Offenders: A Randomized Controlled Trial
Brief Title: Omega-3 Supplements to Reduce Antisocial Behaviour in Young Offenders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Singapore Prison Service (Other Government)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SingaporePS
Record Dates: First submitted 2018-07-31; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Antisocial Behavior
MeSH Terms: conditions — Antisocial Personality Disorder | interventions — Docosahexaenoic Acids; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Omega-3 (Experimental): this group receives a fruit juice drink containing omega-3
  Interventions: Combination Product: Omega-3; Other: Treatment as Usual
- Placebo (Placebo Comparator): this group receives the same fruit juice drink as in the experimental group, but it does not contain omega-3
  Interventions: Combination Product: Placebo; Other: Treatment as Usual
- Treatment as Usual (Other): this group do not receive a fruit juice drink
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Combination Product: Omega-3 — 1g of omega-3 supplement to be taken per day for a duration of 3 months in the form of a fruit juice drink
  Arms: Omega-3
Combination Product: Placebo — Fruit juice drink only
  Arms: Placebo
Other: Treatment as Usual — Young Offenders Intervention Programme

SUMMARY:
The study aims to examine the effects of providing omega-3 supplements on young offenders' antisocial behaviour. Participants will be randomized into three groups: (1) Omega-3, (2) Placebo and (3) Treatment as Usual. Self report and correctional officer ratings of behaviour will be assessed at 0 months (baseline), 3 months (end of supplementation), 6 months and 12 months. The investigators hypothesize that omega-3 supplementation will reduce antisocial behaviour among the young offenders.

DETAILED DESCRIPTION:
This study follows up on two prior omega-3 supplementation Randomized Controlled Trial (RCT) conducted on young offenders - one in the UK (Gesch et al. 2002) and the Netherlands (Zaalberg et al. 2009).

ELIGIBILITY:
Inclusion Criteria:

* Admission into young offender's institution

Exclusion Criteria:

* Allergy to fish and fish products
* Serious mental illness and intellectual disability
* Ability to read and write at the level required to complete self report questionnaires

Ages: 16 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 181 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2013-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Antisocial Behaviour (Aggression) at 3 months, 6 months and 12 months | 0 Months (baseline), 3 Months, 6 Months, 12 Months
  Proactive and Reactive Aggression Questionnaire (23 items). Scale of 0 (Never), 1 (Sometimes) and 2 (Often). Total range: 0 (min) to 46 (max). Higher scores indicate higher levels of aggression. 2 subscales: proactive aggression (range: 0 to 22) and reactive aggression (range: 0 to 22). Total and subscale scores computed by summing up the respective items.
Change in Antisocial Behaviour (Conduct and Oppositional Defiance) at 3 months, 6 months and 12 months | 0 Months (baseline), 3 Months, 6 Months, 12 Months
  Conduct and Oppositional Defiant Disorder Questionnaire (20 items). Scale of 0 (Never), 1 (Sometimes) and 2 (Often). Total range: 0 (min) to 40 (max). Higher scores indicate higher levels of Oppositional Defiant Disorder, Conduct Disorder and antisocial behaviour. 2 subscales: Oppositional Defiant Disorder (range: 0 to 16),Conduct Disorder (range: 0 to 24). Total and subscale scores are computed by summing up the respective items.

SECONDARY OUTCOMES:
Schizotypal Personality | 0 Months (baseline), 3 Months, 6 Months, 12 Months
  Schizotypal Personality Questionnaire - Brief. The questionnaire consist of 22 items, with participants providing responses in a binary (Yes / No) format. "Yes" is scored as a 1, while "No" is scored a 0, therefore the scale ranges from 0 (min) to 22 (max). Higher scores represent greater levels of schizotypal personality pattern. There are three subscales: interpersonal (range: 0 to 8), cognitive perceptual (range: 0 to 8) and disorganized (0 to 6). Both total and subscale scores are computed by summing up the respective items.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Raine, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
Requests for data will be reviewed by the Singapore Prison Service.